CLINICAL TRIAL: NCT04014556
Title: Aflibercept Plus Micropulse Laser Versus Aflibercept Monotherapy for Diabetic Macular Edema. One Year Results of a Randomized Clinical Trial
Brief Title: Aflibercept Plus Micropulse Laser Versus Aflibercept Monotherapy for Diabetic Macular Edema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Mahmoud Abouhussein, Assistant professor, University of Alexandria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 31181
Record Dates: First submitted 2019-07-05; First posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aflibercept plus micropulse laser (group A) (Active Comparator): Overall 40 patients were included in the study; they were randomized into either group A (Aflibercept + Micropulse; 20 patients) or group B (Aflibercept monotherapy; 20 patients).
  Interventions: Device: micropulse laser; Drug: Aflibercept
- Aflibercept monotherapy (group B) (Active Comparator): Overall 40 patients were included in the study; they were randomized into either group A (Aflibercept + Micropulse; 20 patients) or group B (Aflibercept monotherapy; 20 patients).
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Device: micropulse laser — Micropulse session details:
  Mainster focal grid contact lens (×1.05 laser magnification) was used to perform laser. The 577-nm yellow laser (OcuLight SLx, Iridex Corp., Mountain View, California, USA) was used. Fixed treatment parameters were used in all cases: 200-μm spot size, 200-ms exposure duration, 400-mW power, and a 5% duty cycle. Confluent applications with no spacing were administered using 5x5 grid pattern over the entire edematous area including the fovea.
  Arms: Aflibercept plus micropulse laser (group A)
Drug: Aflibercept — Aflibercept

SUMMARY:
Purpose: To evaluate the role of adjuvent micropulse laser with Aflibercept injections in the management of treatment naïve centre involving DME, looking at decreased treatment burden and increased efficacy as outcomes.

Methods: This was a prospective, single centre, randomized trial that included 40 eyes (40 patients) with previously untreated centre involved DME. Patients were randomly assigned to receive either Aflibercept plus micropulse laser (group A) or Aflibercept monotherapy (group B).

DETAILED DESCRIPTION:
Patients were randomly distributed in a 1:1 ratio between the two studied groups. Group A received 3 monthly injections of Aflibercept 2 mg/0.05 mL (Eylea; Bayer, Berlin, Germany) as a loading dose, followed one month later by one 577 nm yellow micropulse laser session with monthly PRN Aflibercept injections. Group B received 3 monthly injections of Aflibercept 2 mg/0.05 mL as a loading dose, followed by monthly PRN Aflibercept injections. Patients in both groups were assessed one month after the end of loading phase; At this point, group A received the micropulse laser session and started PRN Aflibercept injections, while group B started PRN Aflibercept injections without receiving the micropulse laser session. After that, both groups were followed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* patients were older than 18 with the clinical diagnosis of previously untreated centre involved DME documented by fluorescein angiography and central macular thickness (CMT) ≥ 300 µm on the spectral-domain OCT Best corrected visual acuity was better than 3/60 with Hb A1C less than 10%.

Exclusion Criteria:

* any previous treatment for DME, proliferative diabetic retinopathy, macular ischemia on fluorescein angiography, epiretinal membrane or tractional maculopathy on OCT, media opacity and any previous intraocular surgery with the exception of uneventful cataract surgery more than 6 months before the beginning of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
The number of Aflibercept injections in both groups | 12 months
  The number of Aflibercept injections in both groups

SECONDARY OUTCOMES:
The changes in visual acuity in both groups. | 12 months
  best corrected visual acuity in both groups at one year.
The changes in central macular thickness in both groups. | 12 months
  central macular thickness in both groups at one year

IPD SHARING:
Plan to Share IPD: No
patient data protection